CLINICAL TRIAL: NCT02774733
Title: Correlation Between the Pulmonary Function Parameters and the Circulatory Parameters of Retrobulbar Blood Vessels in Patients With Type 2 Diabetes
Brief Title: Correlation Between the Pulmonary Function Parameters and the Circulatory Parameters (PSV, EDV, RI) of Retrobulbar Blood Vessels (CRA, PCA, and OA) in 48 T2DM Patients Did Not Combinate With DR
Acronym: CPCT2DM
Status: Completed | Type: Observational
Sponsor: Fourth People's Hospital of Shenyang (Other)
Responsible Party: Principal Investigator, Jin-song Kuang, Chief physician, Fourth People's Hospital of Shenyang
Other Study IDs: F11-262-9-25
Record Dates: First submitted 2016-05-07; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

INTERVENTIONS:
Device: spirometer;Intraocular pressure;Color doppler imaging

SUMMARY:
Objective: The main target of this study was to research the correlation between the pulmonary function and the circulatory parameters of retrobulbar blood vessels in patients with type 2 diabetes (T2DM) without diabetic retinopathy (DR).

Method: T2DM patients without DR were choose to research the correlation between the pulmonary function and the circulatory parameters of retrobulbar blood vessels. The primary endpoints were the pulmonary function parameters; The secondary endpoints were the HbA1c, FPG, 2hPG, WC, and BMI. The tertiary endpoints were the blood-fat; In addition, the retrobulbar circulation in the retrobulbar blood vessels were evaluated using color doppler imaging (CDI).

DETAILED DESCRIPTION:
Pulmonary function parameters (VC%, FVC%, FEV1%, PEF%, MVV%, TLC%, FEV1/FVC%, DLCO%, and DLCO/VA%); the retrobulbar circulation (PSV, EDV, RI);retrobulbar blood vessels (CRA, PCA, and OA);blood-fat(TC, HDL-C, LDL-C, and TG).

Pulmonary function was measured by spirometer which was provided by Jaska Corporation in Japan, model number: HI-101; The CDI recordings were taken using a Powervision SSA-380A (Toshiba, Japan) using a 7-MHz transducer.

ELIGIBILITY:
Inclusion Criteria:

1. The patients were diagnosed with T2DM according to the guidelines of the American Diabetes Association;
2. No smoking history, pulmonary disease nor pulmonary infection within a fortnight;
3. Did not have hepatopathy, nephropathy, and gastrointestinal disease; and
4. Likely to have good compliance and able to visit our hospital for periodic assessments.

Exclusion Criteria:

1. T1DM, gestation and lactation;
2. Renal inadequacy, a serum creatinine >132 µmol/L (male), or a serum creatinine >123 µmol/L (female);
3. hypohepatia, the liver enzyme was two times higher than normal;
4. Intensive care with insulin treatment;
5. The patients combinated with DR and hypertension (antihypertensive drugs were used);
6. Patients with other eye conditions that could affect the blood flow, such as high degree myopia, maculopathy of any origin, glaucoma, and those with a history of laser treatment or introacular surgery;
7. New York Heart Association class III or IV heart failure, a history of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within 6 months; 8) Cholesterol-lowering drugs can not control the blood-fat (TC > 250 mg/dl, HDL-C < 30 mg/dL, LDL-C > 170 mg/dl, TG > 200 mg/dl) adequately; and

9) Use of systemically injected glucocorticoids within 3 months prior to our study.

Ages: 34 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Investigators selected 60 patients (34 males, 26 females) with T2DM from the the diabetic outpatient clinic in Shenyang the Fourth Hospital of People, but only 48 patients (26 males, 22 females) can be researched in our study. All patients were provided a diet and exercise program by professional nutritionists. The race ratio (all were Chinese Hans), age (range from 34 to 68 years), diabetes duration (range from 3 to 12 years), BMI (range from 20 to 30 kg/m2), HbA1c [ range from 7.0 % (53 mmol/mol) to 10 % (86 mmol/mol) ]. Through the detecting, we excluded 6 patients (4 were in A1 stage, 2 was in A2 stage) because of DR. Finally, 48 patients (26 males, 22 females) completed the study.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The pulmonary function (using spirometer)of three categories of patients, based on HbA1c levels, were compared | one week
  pulmonary function parameters include: VC%, FVC%, FEV1%, PEF%, MVV%, TLC%, FEV1/FVC%, DLCO%, and DLCO/VA%;HbA1c levels: ≥ 8.0, < 8.0 and > 7.0, ≤ 7.0
The circulatory parameters (using CDI)of retrobulbar blood vessels of three categories of patients, based on HbA1c levels, were compared | one week
  retrobulbar blood vessels include CRA, PCA, and OA; circulatory parameters include PSV, EDV, and RI; HbA1c levels: ≥ 8.0, < 8.0 and > 7.0, ≤ 7.0
The correlation between the pulmonary function parameters and the retrobulbar circulation parameters in 48 T2DM patients | one week

SECONDARY OUTCOMES:
HbA1c, FPG, 2hPG, WC,BMI, DBP, SBP, and blood-fat in 48 T2DM patients | one week
  blood-fat include TC, HDL-C, LDL-C, and TG

REFERENCES:
- [Derived] Tai H, Wang MY, Zhao YP, Li LB, Jiang XL, Dong Z, Lv XN, Liu J, Dong QY, Liu XG, Kuang JS. Pulmonary Function and Retrobulbar Hemodynamics in Subjects With Type 2 Diabetes Mellitus. Respir Care. 2017 May;62(5):602-614. doi: 10.4187/respcare.05129. Epub 2017 Feb 28. PMID 28246307